CLINICAL TRIAL: NCT03615235
Title: APOL1 Long-term Kidney Transplantation Outcomes Network (APOLLO)
Acronym: APOLLO
Status: Recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00051561; U01DK116041 (NIH); U01DK116040 (NIH)
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-06

CONDITIONS: Kidney Diseases; Kidney Failure; Kidney Disease, Chronic
Keywords: Apolopoprotein L1 gene (APOL1); Kidney Transplantation; Kidney Donor; United Network for Organ Sharing (UNOS); Association of Organ Procurement Organizations (AOPO); Kidney Transplantation Outcomes Network
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood for DNA extraction, serum, urine, kidney biopsy samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Recipients of a Kidney Transplant: APOLLO will prospectively assess transplant outcomes in recipients of kidneys from eligible living and deceased donors at all transplant programs in the United States including Puerto Rico.
- Living Kidney Donors: APOLLO will prospectively assess post-donation renal outcomes in eligible living kidney donors at all transplant programs in the United States including Puerto Rico.

SUMMARY:
The APOLLO study is being done in an attempt to improve outcomes after kidney transplantation and to improve the safety of living kidney donation based upon variation in the apolipoprotein L1 gene (APOL1). Genes control what is inherited from a family, such as eye color or blood type. Variation in APOL1 can cause kidney disease. African Americans, Afro-Caribbeans, Hispanic Blacks, and Africans are more likely to have the APOL1 gene variants that cause kidney disease. APOLLO will test DNA from kidney donors and recipients of kidney transplants for APOL1 to determine effects on kidney transplant-related outcomes.

DETAILED DESCRIPTION:
The National Institutes of Health (NIH)-sponsored collaborative APOL1 Long-term Kidney Transplantation Outcomes Network (APOLLO) is charged with prospectively assessing the effects of renal-risk variants (RRVs) in the apolipoprotein L1 gene (APOL1) on outcomes for kidneys from donors with recent African ancestry and the recipients of their kidneys, after deceased- and living-donor renal transplantation. For the purposes of APOLLO, recent African ancestry is defined as individuals with similar genetic make-up to those currently residing in Africa. APOLLO will also study the impact of APOL1 RRVs on the health of living kidney donors with recent African ancestry.

ELIGIBILITY:
Inclusion Criteria for Living Donors:

* Living kidney donors with self-reported recent African ancestry (defined as African American, Afro-Caribbean, Hispanic black or African) will be eligible for inclusion.

Exclusion Criteria for Living Donors:

* Participants who are unable or unwilling to provide informed consent.

Enrollment and bio sample collection from deceased donors at OPOs ended on May 31, 2023 and recruiting kidney transplant recipients ended on June 15, 2023.

Phase II started on 9/1/2023 and only Living Donors will be recruited for an additional 2 years.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Thirteen APOLLO Clinical Centers (CCs) will prospectively enroll eligible living kidney donors and recipients of kidney transplants from eligible living and deceased kidney donors at all transplant programs in the continental United States including Puerto Rico. The APOLLO Scientific and Data Research Center (SDRC or Coordinating Center) will support and participate in studies determining the impact of donor and recipient APOL1 genotypes on kidney transplant outcomes in recipients of a kidney transplant from a donor with recent African ancestry, and follow African ancestry living kidney donors for changes in vital status, kidney function and proteinuria. In this protocol, recent African ancestry is broadly defined as African American, Afro-Caribbean, Hispanic black, and African.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-03-21 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Time to death-censored renal allograft failure from the UNOS database | up to 4.5 years
  Time from receipt of kidney transplant to death-censored renal allograft failure. Measured in days.

SECONDARY OUTCOMES:
The rate of loss of renal clearance function from clinical laboratory data | up to 4.5 years
  Rate of change in the estimated glomerular filtration rate Measured in ml/min/1.73 m2.
The rate of change in serum creatinine concentration from clinical laboratory data | up to 4.5 years
  Rate of change in the reciprocal of the serum creatinine concentration. Measured as 1/serum creatinine concentration [in mg/dl].
Time to sustained development of overt proteinuria in the outpatient setting. | up to 4.5 years
  Overt proteinuria is defined as urine protein:creatinine ratio (UPCR) >500 mg/g, urine albumin:creatinine ratio (UACR) >300 mg/g, or >2+ proteinuria on urine dipstick. This outcome requires repeat documentation of proteinuria using either UPCR, UACR or dipstick test >1 month after initial detection based on clinic data
Rate of change in kidney function and quantitative proteinuria from baseline pre-donation levels in living kidney donors (to include effects on stages of CKD) | up to 4.5 years
  Rate of change (i.e., slope of change) in estimated glomerular filtration rate based on serum creatinine concentration from UNOS and clinic data
Renal allograft failure in patients with End Stage Renal Disease defined based on Standardized Outcomes in Nephrology (SONG) criteria | up to 4.5 years
  Renal allograft failure in patients with End Stage Renal Disease defined based on Standardized Outcomes in Nephrology (SONG) criteria: return to chronic renal replacement therapy (dialysis for >90 days or submission of Centers for Medicare and Medicaid Services End Stage Renal Disease Medical Evidence Report [2728 Form]) or repeat kidney transplantation.36 This definition of renal allograft failure specifically excludes acute kidney injury (AKI), delayed graft function (DGF), or primary non-function (requirement of dialysis for the initial 90 days after kidney transplant or re-transplant within 90 days). The diagnoses of AKI, DGF and primary non-function will be abstracted from UNOS, clinic notes and hospital discharge summaries.
The effects of donor APOL1 RRVs on time to "death or renal allograft failure" using UNOS data for all recipients of an APOLLO Deceased Donor Kidney Transplant. | up to 4.5 years
  The effects of donor APOL1 RRVs on time to "death or renal allograft failure" using UNOS data for all recipients of an APOLLO Deceased Donor Kidney Transplant.
he effects of donor APOL1 RRVs on time to "death-censored renal allograft failure (using UNOS data) or death from Corona Virus Disease of 2019 infection (COVID-19) | up to 4.5 years
  The effects of donor APOL1 RRVs on time to "death-censored renal allograft failure (using UNOS data) or death from Corona Virus Disease of 2019 infection (COVID-19) (using APOLLO transplant program data)" among the subset of consented recipients of an APOLLO Deceased Donor Kidney Transplant

CONTACTS AND LOCATIONS:
Overall Officials: Barry I. Freedman, MD, Principal Investigator — Wake Forest University Health Sciences; David M. Reboussin, PhD, Principal Investigator — Wake Forest University Health Sciences; Paul L. Kimmel, MD, Study Director — Natl Institute of Diabetes, Digestive & Kidney Diseases; Marva Moxey-Mims, MD, Study Chair — Children's Natl Health System; George Washington Univ Sch of Med and Health Serv
Locations (18):
- United States (18):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California San Francisco, San Francisco, California
  - University of Miami / Miami Transplant Institute, Miami, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Joslin Diabetes Center / Harvard University, Boston, Massachusetts
  - University of Michigan Medicine, Ann Arbor, Michigan
  - Saint Louis University Center for Transplantation, St Louis, Missouri
  - Ichan School of Medicine at Mount Sinai, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Duke University, Durham, North Carolina
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Wisconsin - Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Study participants will have the option of receiving their APOL1 genotype test result from a Clinical Laboratory Improvement Amendments (CLIA) research lab. Deceased donor family decision makers will also have the option of receiving their loved one's APOL1 genotype test result from a CLIA research lab. Results will be made available after enrollment is complete.Those who wish to receive these results will have been informed of benefits and risks of requesting and receiving this information prior to consenting to participate in APOLLO and again at the time of requesting test results. Info graphics to aid in the decision process for requesting Individual Participant Data (IPD) are provided at the time of consent and on the APOLLO website. Prior to sending IPD, participants and deceased donor family decision makers will be asked to verify that they received and understand the information. They will be able to ask questions to local study staff or the Coordinating Center.
Supporting Information: ICF
Time Frame: Approximately 3 years after enrollment begins (once all testing is performed at once). Results will be available for 12 months.
Access Criteria: Requests for return of IPD will be made via the APOLLO website. Individual letters containing IPD and explanations of results will come via the United States Postal Service.
URL: http://TheApolloNetwork.org

REFERENCES:
- [Background] Freedman BI, Moxey-Mims M. The APOL1 Long-Term Kidney Transplantation Outcomes Network-APOLLO. Clin J Am Soc Nephrol. 2018 Jun 7;13(6):940-942. doi: 10.2215/CJN.01510218. Epub 2018 Apr 27. No abstract available. PMID 29703792
- [Background] Freedman BI, Julian BA. Evaluation of Potential Living Kidney Donors in the APOL1 Era. J Am Soc Nephrol. 2018 Apr;29(4):1079-1081. doi: 10.1681/ASN.2018020137. Epub 2018 Mar 9. No abstract available. PMID 29523593
- [Background] Freedman BI, Locke JE, Reeves-Daniel AM, Julian BA. Apolipoprotein L1 Gene Effects on Kidney Transplantation. Semin Nephrol. 2017 Nov;37(6):530-537. doi: 10.1016/j.semnephrol.2017.07.006. PMID 29110760
- [Background] Julian BA, Gaston RS, Brown WM, Reeves-Daniel AM, Israni AK, Schladt DP, Pastan SO, Mohan S, Freedman BI, Divers J. Effect of Replacing Race With Apolipoprotein L1 Genotype in Calculation of Kidney Donor Risk Index. Am J Transplant. 2017 Jun;17(6):1540-1548. doi: 10.1111/ajt.14113. Epub 2017 Jan 3. PMID 27862962
- [Background] Dorr CR, Freedman BI, Hicks PJ, Brown WM, Russell GB, Julian BA, Pastan SO, Gautreaux MD, Muthusamy A, Chinnakotla S, Hauptfeld V, Bray RA, Kirk AD, Divers J, Israni AK. Deceased-Donor Apolipoprotein L1 Renal-Risk Variants Have Minimal Effects on Liver Transplant Outcomes. PLoS One. 2016 Apr 7;11(4):e0152775. doi: 10.1371/journal.pone.0152775. eCollection 2016. PMID 27054572
- [Background] Freedman BI, Pastan SO, Israni AK, Schladt D, Julian BA, Gautreaux MD, Hauptfeld V, Bray RA, Gebel HM, Kirk AD, Gaston RS, Rogers J, Farney AC, Orlando G, Stratta RJ, Mohan S, Ma L, Langefeld CD, Bowden DW, Hicks PJ, Palmer ND, Palanisamy A, Reeves-Daniel AM, Brown WM, Divers J. APOL1 Genotype and Kidney Transplantation Outcomes From Deceased African American Donors. Transplantation. 2016 Jan;100(1):194-202. doi: 10.1097/TP.0000000000000969. PMID 26566060
- [Background] Freedman BI, Julian BA. Should kidney donors be genotyped for APOL1 risk alleles? Kidney Int. 2015 Apr;87(4):671-3. doi: 10.1038/ki.2015.16. No abstract available. PMID 25826538
- [Background] Freedman BI, Julian BA, Pastan SO, Israni AK, Schladt D, Gautreaux MD, Hauptfeld V, Bray RA, Gebel HM, Kirk AD, Gaston RS, Rogers J, Farney AC, Orlando G, Stratta RJ, Mohan S, Ma L, Langefeld CD, Hicks PJ, Palmer ND, Adams PL, Palanisamy A, Reeves-Daniel AM, Divers J. Apolipoprotein L1 gene variants in deceased organ donors are associated with renal allograft failure. Am J Transplant. 2015 Jun;15(6):1615-22. doi: 10.1111/ajt.13223. Epub 2015 Mar 24. PMID 25809272
- [Background] Reeves-Daniel AM, DePalma JA, Bleyer AJ, Rocco MV, Murea M, Adams PL, Langefeld CD, Bowden DW, Hicks PJ, Stratta RJ, Lin JJ, Kiger DF, Gautreaux MD, Divers J, Freedman BI. The APOL1 gene and allograft survival after kidney transplantation. Am J Transplant. 2011 May;11(5):1025-30. doi: 10.1111/j.1600-6143.2011.03513.x. Epub 2011 Apr 12. PMID 21486385
- [Background] Lee BT, Kumar V, Williams TA, Abdi R, Bernhardy A, Dyer C, Conte S, Genovese G, Ross MD, Friedman DJ, Gaston R, Milford E, Pollak MR, Chandraker A. The APOL1 genotype of African American kidney transplant recipients does not impact 5-year allograft survival. Am J Transplant. 2012 Jul;12(7):1924-8. doi: 10.1111/j.1600-6143.2012.04033.x. Epub 2012 Apr 4. PMID 22487534
- [Background] Doshi MD, Ortigosa-Goggins M, Garg AX, Li L, Poggio ED, Winkler CA, Kopp JB. APOL1 Genotype and Renal Function of Black Living Donors. J Am Soc Nephrol. 2018 Apr;29(4):1309-1316. doi: 10.1681/ASN.2017060658. Epub 2018 Jan 16. PMID 29339549